CLINICAL TRIAL: NCT04643756
Title: Investigation of the Effects of Two Different Treatment Programs on Pain Severity, Low Back Awareness, Functional and Psychosocial Factors in Patients With Chronic Low Back Pain
Brief Title: Investigation of the Effects of Two Different Treatment Programs on Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Özgür Nadiye Karaman, Physiotherapist, MSc, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 60116787-020/62195
Record Dates: First submitted 2020-11-05; First posted 2020-11-25 (Actual); Last update posted 2021-09-13 (Actual); Status verified 2021-09

CONDITIONS: Chronic Low-back Pain
Keywords: chronic low back pain, kinesiotape, physiotherapy, awareness

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Physiotherapy (Active Comparator): Classical electrotherapy method consisting of tens, hotpack and ultrasound. Procedure/Device: Conventional Physiotherapy Conventional Physiotherapy consist of Hotpacks, TENS and US.The participants were positioned in prone and supported with a pillow under the abdomen, 20 min hot pack was applied. Therapatic Ultrason were applied with the frequency of 1 MHz, intensity of 1,5 watt/cm2 and duration of 5 minute. TENS was applied to the lumbar region with 2-channel, 4 surface electrodes at 60-120 Hz, and 50-100 pulse duration for 20 minutes.
  Interventions: Other: conventional physiotherapy
- Conventional Physiotherapy + Kinesiotaping (Active Comparator): Kinesiotaping application in addition to classical electrotherapy method consisting of tens, hotpack and ultrasound.It will be applied to reduce pain, increase proprioception and awareness. Kinesiotaping will be re-applicated every day. Space taping will be applied to the waist area. Space taping creates a vacuum effect on the skin, loosening the adhesions in the tissue layers. With this lifting effect, it creates a space under the skin, causing an increase in circulation and a decrease in pain. Four pieces of I-tape will be used for taping. The middle point of the first tape will be attached with maximum tension. The ends of the tape will be tensionless. The second tape will also be applied at a 90 degree angle. The third and fourth tapes will be taped at an angle of 45 degrees.
  Interventions: Other: conventional physiotherapy plus kinesiotaping

INTERVENTIONS:
Other: conventional physiotherapy — Classical electrotherapy method consisting of tens, hotpack and ultrasound.
  Arms: Conventional Physiotherapy
Other: conventional physiotherapy plus kinesiotaping — Conventional physiotherapy plus kinesiotaping
  Arms: Conventional Physiotherapy + Kinesiotaping

SUMMARY:
This study was planned to examine the effects of two different treatment programs on pain intensity, back awareness, functional and psychosocial factors in patients with chronic low back pain.

DETAILED DESCRIPTION:
Recent study will be carried out on volunteer patients who applied to the Physical Therapy Clinic of "Mugla Sitki Kocman University" Training and Research Hospital, who were diagnosed with chronic non-specific low back pain and who comply with the study criteria.

The sample size has been calculated that 80% power can be obtained at 95% confidence level. It was found that at least 21 cases, a total of 44 cases, were required for each group.

Volunteers will be divided into 2 groups by randomization. Conventional physiotherapy applications will be applied to the control group. In addition to conventional physiotherapy methods, kinesio-taping (KT) will be applied to the study group. Patients in both groups will be treated 5 days a week for a total of 10 sessions for 2 weeks. KT will be renewed in each session on weekdays.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged 18 to 60 years with chronic low back pain
* Those who have complained of low back pain for at least 3 months
* Individuals whose pain intensity is above 3.5 cm according to VAS
* Pain and numbness that does not spread to the legs

Exclusion Criteria:

* Situations that prevent the evaluation or communication with the individual
* Illiterate individuals
* Individuals who have undergone surgical operations on the spine and / or extremities
* Conditions where specific pathological conditions are proven such as malignant condition, fracture, systemic rheumatoid disease
* Orthopedic and neurological problems that prevent evaluation and / or treatment
* Complaints of pain and numbness spreading to the lower extremities
* Individuals with a diagnosed psychiatric illness
* Individuals who have received physiotherapy in the last 6 months
* Individuals who use another treatment method during the study
* Individuals with musculoskeletal pain in any other part of the body during work
* Pregnant

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
Pain assessment Change from baseline at 3 weeks and Change from baseline at 6 weeks | Baseline, 3 weeks, 6 weeks
  Visual Analogue Scale (VAS): The patient is asked to mark the pain felt on a 10 cm.
Awareness Assessment Change from baseline at 3 weeks and Change from baseline at 6 weeks | Baseline, 3 weeks, 6 weeks
  Fremantle Back Awareness Questionnaire (FreBAQ): FreBAQwill be used for awareness.
Functional assessment Change from baseline at 3 weeks and Change from baseline at 6 weeks | Baseline, 3 weeks, 6 weeks
  Repeated Sit-to-Stand Test
Assessment of depression and anxiety level Change from baseline at 3 weeks and Change from baseline at 6 weekschanging from baseline at 6 weeks | Baseline, 3 weeks, 6 weeks
  Hospital and Anxiety Depression Scale (HADS):Anxiety and depression levels will be evaluated subjectively with the Hospital Anxiety and Depression Scale.
Assessing Kinesophobia Change from baseline at 3 weeks and Change from baseline at 6 weeks | Baseline, 3 weeks, 6 weeks
  Fear-Avoidance Beliefs Questionnaire (FABQ):It measures the patient's fear of movement caused by low back pain.
Timed Up and Go Test Change from baseline at 3 weeks and Change from baseline at 6 weeks | Baseline, 3 weeks, 6 weeks
  Timed Up and Go Test
Modified Schober Test Change from baseline at 3 weeks and Change from baseline at 6 weeks | Baseline, 3 weeks, 6 weeks
  Modified Schober Test
Disability level Change from baseline at 3 weeks and Change from baseline at 6 weeks. | Baseline, 3 weeks, 6 weeks
  Roland Morris Disability Questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Emine PT Aslan Telci, Prof. Dr, Study Director — Pamukkale University
Locations (1):
- Emine Aslan Telci, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nelson NL. Kinesio taping for chronic low back pain: A systematic review. J Bodyw Mov Ther. 2016 Jul;20(3):672-81. doi: 10.1016/j.jbmt.2016.04.018. Epub 2016 Apr 27. PMID 27634093
- [Background] Paoloni M, Bernetti A, Fratocchi G, Mangone M, Parrinello L, Del Pilar Cooper M, Sesto L, Di Sante L, Santilli V. Kinesio Taping applied to lumbar muscles influences clinical and electromyographic characteristics in chronic low back pain patients. Eur J Phys Rehabil Med. 2011 Jun;47(2):237-44. Epub 2011 Mar 24. PMID 21430611
- [Background] Kachanathu SJ, Alenazi AM, Seif HE, Hafez AR, Alroumim MA. Comparison between Kinesio Taping and a Traditional Physical Therapy Program in Treatment of Nonspecific Low Back Pain. J Phys Ther Sci. 2014 Aug;26(8):1185-8. doi: 10.1589/jpts.26.1185. Epub 2014 Aug 30. PMID 25202177
- [Result] Li Y, Yin Y, Jia G, Chen H, Yu L, Wu D. Effects of kinesiotape on pain and disability in individuals with chronic low back pain: a systematic review and meta-analysis of randomized controlled trials. Clin Rehabil. 2019 Apr;33(4):596-606. doi: 10.1177/0269215518817804. Epub 2018 Dec 11. PMID 30526011